CLINICAL TRIAL: NCT02270216
Title: Study of Cardiovascular Responses to Static and Dynamic Exercise in Isolated Systolic Hypertension
Brief Title: Cardiovascular Responses to Static and Dynamic Exercise in Elderly With Isolated Systolic Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sahachat Aueyingsak (Other)
Responsible Party: Sponsor-Investigator, Sahachat Aueyingsak, Master's Degree Student, Khon Kaen University
Organization: Khon Kaen University (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: KhonKaenU
Record Dates: First submitted 2014-10-14; First posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Cardiovascular Responses in Elderly With Isolated Systolic Hypertension
Keywords: isolated systolic hypertension; exercise pressor responses
MeSH Terms: conditions — Isolated Systolic Hypertension | interventions — Exercise

ARMS (2):
- elderly with isolated systolic hypertension (Active Comparator): over 60 years of age with essential isolated systolic hypertension (stage I-II base on recommendation of JNC-VII) for the hypertension group. Good communication, independent physical activity. The healthy subject should be non-smokers, free of any signs or symptoms of disease as revealed by medical history
  Interventions: Procedure: static hand grip exercise; Procedure: cycling exercise
- healthy elderly (Active Comparator): over 60 years of age with normal blood pressure in the healthy group. Good communication, independent physical activity. The healthy subject should be non-smokers, free of any signs or symptoms of disease as revealed by medical history
  Interventions: Procedure: static hand grip exercise; Procedure: cycling exercise

INTERVENTIONS:
Procedure: static hand grip exercise — The static exercise pressor response will be tested using isometric handgrip of the left hand. The forearm will be supported on an arm rest with elbow flexed. The maximum voluntary contraction force will be measured as the best of three attempts. After 2 minute rest, subjects will perform 2 minute of isometric hand grip contraction at 30% MVC. Circulatory occlusion(50 mmHg supra-systolic pressure) will start at 1.30 min and continued for 2 minute after the end of the isometric handgrip exercise. Following release of the cuff there will be a further 2 minutes recovery. The blood pressure and heart rate will be measured at the end of each minute during rest, isometric handgrip, circulatory occlusion and recovery. Subjects will be instructed to breathe normally during the test and avoid any Valsalva maneuver; breathing frequency will be monitored during the handgrip pressor test using capnography.
  Other Names: static exercise
Procedure: cycling exercise — The dynamic exercise will be with the subject sitting on a cycle ergometer (Monark 828 E). Resting heart rate will be measured for 2 minutes before the start of exercise. The exercise level will be limited to 50% of the estimated maximum heart rate reserve. Maximum heart rate will be estimated as 207-0.7*age and heart rate reserve (HRR) as maximum minus resting heart rate. Subjects will pedal at 50 rpm for 1 min with no load and then 3 minutes against a load of 0.5 Kp (25W) increasing to a load of 1 Kp for the next 3 minutes and to 1.5 Kp, if necessary, for a further 3 minutes until the target heart rate of 50% HRR is reached.
  Subjects will be asked about their level of perception of dyspnea using a visual analog scale every 3 minutes at the end of each load. At the end of the exercise, the subjects will sit for ten minutes.

SUMMARY:
Aim to study the exercise responses to both static and dynamic exercise in elderly people with and without essential isolated systolic hypertension, seeking to identify potentially dangerously high responses

DETAILED DESCRIPTION:
1. Design The proposed study is of a experimental study design. The study will be subject to approval by the Ethical committee of Khon Kaen University and subjects will be asked to give their written agreement to participate.
2. Subjects Elderly subjects with isolated systolic hypertension will be recruited from primary care units in the community and outpatient department of Srinakarind hospital in Khon Kaen province. Healthy normotensive subjects living independently with normal physical activity will be recruited from the same community.

   Inclusion criteria: Subjects should be over 60 years of age with essential isolated systolic hypertension (stage I-II base on recommendation of JNC-VII) for the hypertension group and normal blood pressure in the healthy group. Good communication, independent physical activity. The healthy subject should be non-smokers, non-obese, free of any signs or symptoms of disease as revealed by medical history Exclusion criteria: Essential hypertension stage III or secondary hypertension, any history of respiratory disease, heart disease, renal disease, blindness, cerebrovascular disease, exercise limited by pain Subjects who have passed the inclusion criteria and exclusion criteria will undertake a dynamic exercise test and a static hand-grip exercise pressor test in the cardiopulmonary research room , Khon Kaen University
3. Outcome measurements The main outcome measures will be changes in blood pressure and heart rate during the two forms of exercise.

   Blood pressure: Blood pressure will be measured with a digital bedside monitor (Figure 1). An inflatable cuff placed around the subject's arm one inch above the patient's elbow over the brachial artery. Resting blood pressure will be measured in a sitting position after having rested for 15 minutes Heart rate: Heart rate will be measured at rest and during exercise. ECG electrode will be attached in lead II configuration and connected to the BIOPAC system. The heart rate will be determined from the R-R interval with the data analyzed by the BIOPAC system.
4. Procedures and protocol After an interview where they will be informed about the various tests and asked to provide their informed consent, the subjects will undertake two different exercise tests, the order of which will be in a randomized and balanced design. The subjects will be asked not to smoke, take alcohol or caffeinated drinks within 2 hours before testing.

   Cycling exercise: The dynamic exercise will be with the subject sitting on a cycle ergometer (Monark 828 E). Resting heart rate will be measured for 2 minutes before the start of exercise. The exercise level will be limited to 50% of the estimated maximum heart rate reserve. Maximum heart rate will be estimated as 207-0.7*age (Gellish et al., 2007) and heart rate reserve (HRR) as maximum minus resting heart rate. Subjects will pedal at 50 rpm for 1 min with no load and then 3 minutes against a load of 0.5 Kp (25W) increasing to a load of 1 Kp for the next 3 minutes and to 1.5 Kp, if necessary, for a further 3 minutes until the target heart rate of 50% HRR is reached.

   Subjects will be asked about their level of perception of dyspnea using a visual analog scale every 3 minutes at the end of each load.

   Static exercise pressor response: The static exercise pressor response will be tested using isometric handgrip of the left hand. The forearm will be supported on an arm rest with elbow flexed. The maximum voluntary contraction force will be measured as the best of three attempts. After 2 minute rest, subjects will perform 2 minute of isometric hand grip contraction at 30% MVC. Circulatory occlusion(50 mmHg supra-systolic pressure) will start at 1.30 min and continued for 2 minute after the end of the isometric handgrip exercise. Following release of the cuff there will be a further 2 minutes recovery. The blood pressure and heart rate will be measured at the end of each minute during rest, isometric handgrip, circulatory occlusion and recovery. Subjects will be instructed to breathe normally during the test and avoid any Valsalva maneuver; breathing frequency will be monitored during the handgrip pressor test using capnography.
5. Data and statistical analysis Data will be expressed as mean ± SD. Changes of data during and post test from baseline. Will be tested by paired t-test. Significance were set at P<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should be over 60 years of age with essential isolated systolic hypertension (stage I-II base on recommendation of JNC-VII) for the hypertension group and normal blood pressure in the healthy group. Good communication, independent physical activity. The healthy subject should be non-smokers, non-obese, free of any signs or symptoms of disease as revealed by medical history

Exclusion Criteria:

* Essential hypertension stage III or secondary hypertension, any history of respiratory disease, heart disease, renal disease, blindness, cerebrovascular disease, exercise limited by pain

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-05; Primary Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | 6 month
  Blood pressure will be measured with a digital bedside monitor. An inflatable cuff placed around the subject's arm one inch above the patient's elbow over the brachial artery. Resting blood pressure will be measured in a sitting position after having rested for 15 minutes
heart rate | 6 month
  Heart rate will be measured at rest and during exercise. ECG electrode will be attached in lead II configuration and connected to the BIOPAC system. The heart rate will be determined from the R-R interval with the data analyzed by the BIOPAC system.

CONTACTS AND LOCATIONS:
Overall Officials: Chulee Jones, PhD, Study Chair — Faculty of Associated Medical Science, Khon Kaen University
Locations (1):
- Khon Kaen University, Khon Kaen, Changwat Khon Kaen, Thailand

REFERENCES:
- See also: The seventh report of the joint national committee on prevention, Detection, evaluation, and treatment of high blood pressure — http://www.ncbi.nlm.nih.gov/pubmed/14656957
- See also: Update on pathophysiology and treatment of hypertension in the elderly. — http://www.ncbi.nlm.nih.gov/pubmed/21681384
- See also: Exaggerated sympathetic and pressor responses to handgrip exercise in older hypertensive humans: role of the muscle metaboreflex — http://www.ncbi.nlm.nih.gov/pubmed/20802135
- See also: Effect of muscle metaboreflex activation on carotid-cardiac baroreflex function in humans — http://www.ncbi.nlm.nih.gov/pubmed/18326794
- See also: The effectiveness of exercise training in lowering blood pressure: a meta-analysis of randomised controlled trials of 4 weeks or longer — http://www.ncbi.nlm.nih.gov/pubmed/9400906
- See also: Effects of aerobic training on exaggerated blood pressure response to exercise in African-Americans with severe systemic hypertension treated with indapamide +/- verapamil +/- enalapril — http://www.ncbi.nlm.nih.gov/pubmed/9165176
- See also: Aging and arterial stiffness — http://www.ncbi.nlm.nih.gov/pubmed/20962429
- See also: RESPeRATE: nonpharmacological treatment of hypertension. — http://www.ncbi.nlm.nih.gov/pubmed/21285661